CLINICAL TRIAL: NCT02282033
Title: Clinical Evaluation of Safety and Performance of the BackBeat Moderato System
Brief Title: Safety and Performance Study of the Moderato System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BackBeat Medical Inc (Industry)
Collaborators: Massachusetts General Hospital (Other); MLM Medical Labs GmbH (Industry); nabios GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-01
Record Dates: First submitted 2014-10-23; First posted 2014-11-04 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Hypertension Resistant to Conventional Therapy; Bradycardia; Atrioventricular Block
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy; Bradycardia; Atrioventricular Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): This is an unblinded, treatment only study in which each patient serves as his or her own control.
  All patients who meet entry criteria will undergo implantation of the Moderato System. During the first month the pacemaker Performance will be evaluated and an additional 3 month period of treatment for studying the Moderato-HTN therapy effect.
  Interventions: Device: The Moderato System

INTERVENTIONS:
Device: The Moderato System — The BackBeat Moderato System incorporates traditional pacing modes and algorithms to provide pacing support to patients with all conditions currently indicated for dual chamber pacing. In addition, a special pacing algorithm was developed to reduce blood pressure.

SUMMARY:
The purpose of the study is to evaluate the safety and performance of the Moderato System by implanting the Moderato pacemaker in patients who require a dual chamber pacemaker, and who also have hypertension, in order to reduce their blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age
* Subject is indicated for implantation or replacement of a dual chamber permanent pacemaker where no lead extraction is necessary.
* Subject has stable regimen of 2 or more maximally tolerated anti-hypertension medications, which is anticipated to be able to be maintained without changes for 3 months.
* Subject has office systolic blood pressure measurements > 140 mmHg on two separate days within a one week period prior to enrollment, and the average of these two measurements is ≥150 mmHg

Exclusion Criteria:

* Subject has known secondary cause of HTN
* Subject has a history of atrial fibrillation
* Subject has ejection fraction <50%
* Subject has symptoms of heart failure of NYHA Class II or more
* Subject has hypertrophic cardiomyopathy, restrictive cardiomyopathy or interventricular septal thickness ≥15 mm
* Subject is on dialysis
* Subject has estimated Glomerular Filtration Rate (GFR) <30 ml/min/1.73m2
* Subject has prior neurological events (stroke or TIA) or carotid artery disease
* Subject has known autonomic dysfunction
* Subject has a history of clinically significant tachyarrhythmia
* Subject has had previous active device-based treatment for hypertension
* Subject has an existing implant, other than a pacemaker that needs replacing
* Subject with average Systolic BP >190 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Moderato Pacing Performance as evaluated through analysis of 24 hour Holter monitoring recordings | 4 months
Moderato Pacing Safety as measured by incidence of of peri-procedural device and treatment-related serious adverse events. | 4 months
  The pacemaker function of the system will be considered to be safe if the rate and severity of pacemaker-related complications is not greater than reported in the literature for similar devices.
Hypertension Treatment Phase Performance as evaluated through analysis of 24 hour Holter monitoring recordings and 24h ambulatory blood pressure. | 3 months
  Moderato - Hypertension device performance will be evaluated through analysis of 24 hour Holter monitoring recordings.
  The device will be considered to be efficacious if there is a reduction of average office blood pressure and/or a reduction in averaged mean 24-hour ambulatory blood pressure.
Hypertension Treatment Phase Safety as measured by Incidence of device- and treatment-related serious adverse events through 3 months of treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Kuck, Prof., Principal Investigator — Asklepios Klinik St. Georg
Locations (10):
- Austria (2):
  - Krankenhaus der Elisabethinen, Linz
  - Medical University Vienna, Vienna
- Chile (2):
  - Clinica Tabancura, Santiago
  - Hospital Dr. Sotero del Rio, Santiago
- Na Homolce Hospital, Prague, Czechia
- Semmelweis University Heart and Vascular Center, Budapest, Hungary
- P. Stradins Clinical University Hospital, Riga, Latvia
- Vilnius University Hospital Santariskiu Klinikos, Vilnius, Lithuania
- Netherlands (2):
  - Academic Medical Center - University of Amsterdam, Amsterdam
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Background] Neuzil P, Merkely B, Erglis A, Marinskis G, de Groot JR, Schmidinger H, Rodriguez Venegas M, Voskuil M, Sturmberger T, Petru J, Jongejan N, Aichinger J, Kamzola G, Aidietis A, Geller L, Mraz T, Osztheimer I, Mika Y, Evans S, Burkhoff D, Kuck KH; BackBeat Study Investigators. Pacemaker-Mediated Programmable Hypertension Control Therapy. J Am Heart Assoc. 2017 Dec 23;6(12):e006974. doi: 10.1161/JAHA.117.006974. PMID 29275370
- See also: Article describing study results — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5779015/